CLINICAL TRIAL: NCT01943916
Title: A Study of Imaging With Opto-acoustics to Diagnose Breast Masses Detected by Mammography and/or Diagnostic Ultrasound: A New Evaluation Tool for Radiologists
Brief Title: The PIONEER-01 Study of the Imagio Breast Imaging System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seno Medical Instruments Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PIONEER-01; NCT01937962 (obsolete NCT alias)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2021-05-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer
Keywords: breast imaging diagnosis; breast ultrasound; Imagio; Seno Medical Instruments, Inc.; Seno; opto-acoustics; OA; angiogenesis; blood map
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imagio OA/US (US and OA/US) (Experimental): Imagio OA/US (gray scale and opto-acoustic)
  Interventions: Device: Imagio OA/US (US and OA/US)
- Imagio gray scale ultrasound (Experimental): Imagio gray scale ultrasound alone
  Interventions: Device: Imagio gray scale ultrasound

INTERVENTIONS:
Device: Imagio OA/US (US and OA/US) — opto-acoustic plus gray scale ultrasound
  Arms: Imagio OA/US (US and OA/US)
Device: Imagio gray scale ultrasound — gray scale ultrasound alone
  Arms: Imagio gray scale ultrasound

SUMMARY:
This is a prospective controlled multi-center study involving gray scale (B-mode) ultrasound vs OA/US (opto-acoustic and gray scale ultrasound) for the visualization of suspicious masses. Imagio gray scale and OA image sets will be collected on each enrolled mass and pushed to an Imaging Core Lab for processing and then to a set of Independent Readers who will read the Imagio gray-scale images vs the Imagio OA/US images.

DETAILED DESCRIPTION:
Imagio is a multi-modality device, comprised of one probe with the ability to image with diagnostic gray scale (B mode) ultrasound alone and gray scale in conjunction with OA together in a six up image.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18 years of age or older
* suspicious mass of breast, identified by a health care practitioner within the past 30 days with diagnostic methodology other than conventional ultrasound.

Exclusion Criteria:

* presence of a condition or impediment that may interfere with imaging.
* pregnant or lactating
* undergoing neoadjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2105 (Actual)
Dates: Start 2012-12-21 (Actual); Primary Completion 2015-09-09 (Actual); Study Completion 2015-09-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Radnet (Temecula), Murrieta, California
  - Sally Jobe, Englewood, Colorado
  - Yale University, New Haven, Connecticut
  - Georgetown University Hospital, Department of Radiology, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Breast Care Atlanta, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - New York Presbyterian Hospital, New York, New York
  - Elizabeth Wende Breast Care, Rochester, New York
  - Solis Women's Health (North Carolina), Greensboro, North Carolina
  - Cleveland Clinic, Breast Services DDI Clinical Research, Cleveland, Ohio
  - Weinstein Imaging Associates, Pittsburgh, Pennsylvania
  - Austin Radiological Association, Austin, Texas
  - MD Anderson Cancer Center, Department of Radiology and Breast Imaging, Houston, Texas
  - Solis Women's Health, Plano, Texas
  - Univ. Texas Health Science Center at San Antontio, Breast Imaging Center at the Cancer Therapy Research Center, San Antonio, Texas

REFERENCES:
- [Background] Otto P, Kist K, Dornbluth NC, McCorvey BM, Zalev J, Herzog D, Clingman B, Miller T, Ermilov S, Nadvoretsky V, Conjusteau A, Su R, Oraevsky A. Clinical Feasibility Study of Combined Opto-Acoustic and Ultrasonic Imaging Modality Providing Co-registered Functional and Anatomical Maps of Breast Tumors. Presented at: 97th Scientific Assembly and Annual Meeting of The Radiological Society of North America; 2011 Nov 28; Chicago, IL.
- [Background] Otto P, Kist K, Dornbluth NC, Herzog D, Clingman B, Ermilov S, Nadvoretsky V, Conjusteau A, Su R, Oraevsky A. Clinical feasibility of Co-registered Opto-acoustic and Ultrasonic Imaging for Differentiation of Breast Tumors. Presented at: Annual Meeting: Society for Nuclear Medicine; 2011 Jun 6; San Antonio, TX.
- [Background] Zalev J (Ryerson Univ, Toronto, Canada), Kolios MC. Detecting Abnormal Vasculature from Photoacoustic Signals Using Wavelet-packet Features. Poster presented at: SPIE Photonics West Symposium; 2011 Jan 22-27; San Francisco, CA.
- [Background] Otto P, Kist K, Dornbluth NC, McCorvey BM, Zalev J, Herzog D, Clingman B, Miller T, Smith R, Ermilov S, Nadvoretsky V, Conjusteau A, Su R, Hernandez T, Oraevsky A. Feasibility of Co-registered Opto-Acoustic and Ulatrsonic Imaging for Differentiation of Malignant from Benign Breast Tumors. Presented at: American Institute of Ultrasound in Medicine Annual Convention; 2012 March 31; Phoenix, AZ.
- [Background] Zalev J, Herzog D, Clingman B, Miller T, Ermilov S, Nadvoretsky V, Conjusteau A, Su R, Tsyboulski D, Oraevsky A, Otto P, Kist K, Dornbluth NC, McCorvey BM. Clinical Feasibility Study of Combined Opto-Acoustic and Ultrasonic Imaging Modality Providing Coregistered Functional and Anatomical Maps of Breast Tumors. Presented at: Photons plus Ultrasound: Imaging and Sensing. SPIE/Bios, Photonics West Symposium; 2012 Jan 22; San Francisco, CA.
- [Background] Otto P, Kist K, Dornbluth NC, McCorvey BM, Miller T, Herzog D, Clingman B, Zalev J, Ermilov S, Oraevsky A. Improve Differentiation of Breast Tumors Using Laser Opto-Acoustic Ultrasonic Imaging System. Poster presented at: European Congress of Radiology; 2012 Mar 1-5; Vienna, Austria.
- [Background] Otto P, Kist K, Dornbluth C, Stavros T, Ulissey M, Herzog D, Clingman B, Zalev J, Lavin P, Oraevsky A. Functional Images of Hemoglobin and Blood Oxygen Saturation Co-registered with Ultrasound Provide Accurate Differentiation of Breast Tumors. Presented at: American Institute of Ultrasound in Medicine Annual Convention; 2013 Apr 6-10; New York, NY.
- [Background] Stavros T, Lerner A, Burak W, Fine R, Boyd B, Miller T, Herzog D, Clingman B, Smith R, Zalev J, Ulissey M. Combining B-Mode Ultrasound and Opto-Acoustic Imaging to Evaluate Breast Lesions. Poster presented at: American Society of Breast Surgeons Annual Meeting; 2013 May 1-5; Chicago, IL.
- [Background] Otto P, Kist K, Dornbluth C, Stavros T, Ulissey M, Herzog D, Clingman B, Zalev J, Lavin P, Oraevsky A. Improved Differentiation of Breast Tumors using Novel Imaging System based on Co-Registered Opto-Acoustic Tomography and Ultrasound. Presented at European Congress of Radiology; 2013 Mar 7-11; Vienna, Austria.
- [Background] Stavros T, Lerner A, Burak W, Fine R, Boyd B, Miller T, Herzog D, Clingman B, Smith R, Zalev J, Ulissey M. Opto-Acoustic Breast Imaging, A New Technology. Poster presented at 23rd Annual National Interdisciplinary Breast Center Conference; 2013 Mar 23-27; Las Vegas, NV.
- [Background] Zalev J, Clingman B, Smith R, Herzog D, Miller T, Stavros AT, Ermilov S, Conjusteau A, Tsyboulski D, Oraevsky A, Kist K, Dornbluth C, Otto P. Real-time Opto-acoustic Imaging System for Clinical Assessment of Breast Lesions. Presented at: Photons plus Ultrasound: Imaging and Sensing, SPIE/BiOS, Photonics West Symposium; 3 Feb 2013; San Francisco, CA.
- [Derived] Ozcan BB, Xi Y, Dogan BE. Supplemental Optoacoustic Imaging of Breast Masses: A Cost-Effectiveness Analysis. Acad Radiol. 2024 Jan;31(1):121-130. doi: 10.1016/j.acra.2023.08.042. Epub 2023 Sep 23. PMID 37748954
- See also: Sponsor website — http://www.senomedical.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective controlled multi-center pivotal study of Imagio Breast Imaging System; two imaging modalities (test and control) used on each subject/mass
Pre-assignment Details: Sixteen (16) centers performing Imagio ultrasound alone (IUS) and Imagio optoacoustic/ultrasound imaging (OA/US) to image breast masses, without using OA/US results for diagnosis; study compared results of each imaging modality (IUS vs. OA/US) to detect malignancy (based on biopsy diagnosis or truth panel decision as ground truth)
Groups:
- Overall Population: Each subject served as her own control, with imaging of each mass by both the test Imagio (IUS+OA) and control (IUS only) modalities; therefore baseline data are not broken into each arm - test and control due the numbers being the same for each arm.
Period: Overall Study
Arm/Group | Overall Population
Started | 2105
Completed | 1739
Not Completed | 366
Not completed — Technically invalid images | 10
Not completed — Enrollment Failure | 23
Not completed — Pilot Phase exclusion | 100
Not completed — Quality Assurance Reader Fail | 130
Not completed — Technical Failure | 39
Not completed — Protocol Deviation No Biopsy | 25
Not completed — No Truth Panel Review | 38
Not completed — Protocol Deviation | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Diagnose (ITD)
Groups:
- Overall Population: Each subject served as her own control, with imaging of each mass by both the test and control modalities; therefore baseline data are for overall population only.
Arm/Group | Overall Population
Number analyzed (Participants) | 1739
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1739
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 255
  Not Hispanic or Latino | 1471
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 57
  Native Hawaiian or Other Pacific Islander | 4
  Black or African American | 216
  White | 1372
  More than one race | 81
  Unknown or Not Reported | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1739
Number of Masses [Number; unit: masses] — Masses evaluated by independent readers Population: Each row is a diagnostic subset. The diagnostic subsets sum to the overall number of subjects.
  masses
    Subjects (Benign + TPB): number analyzed (Participants) | 1038
    Subjects (Benign + TPB) | 1038
    Subjects (Cancer): number analyzed (Participants) | 652
    Subjects (Cancer) | 652
    Subjects (Other-TPC,HR): number analyzed (Participants) | 49
    Subjects (Other-TPC,HR) | 49
Mass Diagnosis [Count of Participants; unit: Participants] — Measure Description: Mass diagnosis by biopsy result or Truth Panel decision on benign status
  Participants
    Subjects (Benign+Truth Panel Benign [TPB]) | 1038
    Subjects (Cancer) | 652
    Subjects (Other-Truth Panel Cancer [TPC], high risk [HR]) | 49

OUTCOME MEASURES:

1. Primary Outcome: Specificity Difference Between Imagio Optoacoustic Plus Gray-scale (OA/US) vs Imagio Gray-scale Ultrasound (IUS)
Description: Primary effectiveness endpoint was the difference in specificity for the Imagio OA/US relative to IUS, across all 7 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth)
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-diagnose population
Measure: Mean (99% Confidence Interval); unit: % benign+TPB masses correctly Id'd
Groups:
- Overall Population: Each subject served as her own control, with imaging of each mass by both the test and control modalities. Specificity difference is a single measure for the overall ITD population.
Arm/Group | Overall Population
Number analyzed (Participants) | 1739
% benign+TPB masses correctly Id'd | 14.9 [12.9 to 16.9]

2. Secondary Outcome: Sensitivity Difference Between Imagio Optoacoustic Plus Gray-scale (OA/US) vs Imagio Gray-scale Ultrasound (IUS)
Description: Sensitivity difference for Imagio OA/US Imagio relative to IUS, across all 7 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth)
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-Diagnose Population
Measure: Mean (99% Confidence Interval); unit: % of malignant masses I'd correctly
Groups:
- Overall Population: Each subject served as her own control, with imaging of each mass by both the test and control modalities. Sensitivity difference is a single measure for the overall ITD population.
Arm/Group | Overall Population
Number analyzed (Participants) | 1739
% of malignant masses I'd correctly | -2.7 [-3.7 to -1.6]

3. Secondary Outcome: Specificity for Each Imaging Modality Imagio Optoacoustic Plus Gray-scale OA/US and Imagio Gray-scale Ultrasound (IUS)
Description: Specificity for each imaging modality, Imagio OA/US (Imagio) and IUS, across all 7 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth)
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-diagnose population
Measure: Mean (99% Confidence Interval); unit: % of benign+TPB masses I'd correctly
Groups:
- Imagio Ultrasound (IUS) Gray-scale Ultrasound Imaging of Mass: Imagio Ultrasound (IUS) gray-scale ultrasound imaging of mass
- OA/US: Imagio optoacoustic + gray-scale ultrasound (OA/US) Imaging of Mass
Arm/Group | Imagio Ultrasound (IUS) Gray-scale Ultrasound Imaging of Mass | OA/US
Number analyzed (Participants) | 1739 | 1739
% of benign+TPB masses I'd correctly | 28.1 [25.8 to 30.5] | 43.0 [40.4 to 45.7]

4. Secondary Outcome: Sensitivity for Each Imaging Modality Imagio Optoacoustic Plus Gray-scale (OA/US) and Imagio Gray-scale Ultrasound (IUS)
Description: Sensitivity for each imaging modality, Imagio OA/US and IUS, across all 7 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth)
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-Diagnose Population
Measure: Mean (99% Confidence Interval); unit: Percentage (%) of malignant masses that
Groups:
- Imagio (OA/US): Imagio optoacoustic imaging plus grayscale imaging of mass
Arm/Group | Imagio Ultrasound (IUS) Gray-scale Ultrasound Imaging of Mass | Imagio (OA/US)
Number analyzed (Participants) | 1739 | 1739
Percentage (%) of malignant masses that | 98.6 [97.8 to 99.1] | 96.0 [94.5 to 97.0]

5. Secondary Outcome: Downgrade Benign Masses Imagio Optoacoustic Plus Gray-scale (OA/US) vs Imagio Gray-scale Imaging (IUS)
Description: Percentage of reads where breast mass was downgraded from one BI-RADS (BR) category to a lower BR category on the basis of additional information from the Imagio OA/US imaging modality compared to IUS, includes reads of each of 7 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth). BR categories used in this study: 2, 3, 4a, 4b, 4c, 5
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-Diagnose Population
Measure: Mean (99% Confidence Interval); unit: Percentage of reads
Groups:
- Overall ITD Population: Each subject served as her own control, with imaging of each mass by both the test and control modalities. Downgrades are based on Imagio optoacoustic plus grayscale (OA/US) relative to Imagio grayscale (IUS), thus this is a single measure for the over all ITD population.
Arm/Group | Overall ITD Population
Number analyzed (Participants) | 1739
Percentage of reads | 34.5 [33.1 to 35.9]

6. Secondary Outcome: Upgrade Cancer Masses - Imagio Optoacoustic Plus Gray-scale (OA/US) vs Imagio Gray-scale Imaging (IUS)
Description: Percentage of reads where breast mass was upgraded from one BI-RADS (BR) category to a higher BR category on the basis of additional information from the Imagio optoacoustic plus grayscale (OA/US) imaging modality compared to Imagio grayscale (IUS), includes reads of each of 7 independent readers; both imaging modalities used in each subject (subject as own control); results for each imaging modality compared to biopsy diagnosis or 12-month follow-up ruling of benign as determined by truth panel (ground truth). BR categories used in this study: 2, 3, 4a, 4b, 4c, 5
Time Frame: Baseline to 12 months +/- 30 days follow-up
Population: Intent-to-Diagnose Population
Measure: Mean (99% Confidence Interval); unit: Percentage of reads
Arm/Group | Overall Population
Number analyzed (Participants) | 1739
Percentage of reads | 0.7 [0.4 to 1.0]

ADVERSE EVENTS:
Time Frame: Subjects followed up post-Imagio (OA/US) and IUS imaging until biopsy or until 12 months (+/-) 30 days; includes truth panel decision of no biopsy.
Description: Safety population (N=1972) reflects all subjects who were exposed to the Imagio (OA/US) device, so this is not the same as the Intent-to-Diagnose (ITD) population used for effectiveness analysis (N=1739).
Groups:
- Safety Population: Each subject served as her own control, with imaging of each mass by both the test and control modalities; therefore safety data are for overall safety population only.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/1972
Serious Adverse Events (participants affected / at risk) | 5/1972
Other Adverse Events (participants affected / at risk) | 47/1972
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=1972)
Device breakage (General disorders) | 1 (1) — (Right saline breast implant rupture)
Atrial fibrillation (Cardiac disorders) | 1 (1) — (Atrial fibrillation)
Cardiac failure congestive (Cardiac disorders) | 1 (1) — (Congestive heart failure)
Non-small cell lung cancer Stage I (Respiratory, thoracic and mediastinal disorders) | 1 (1) — (Stage I, non-small cell lung cancer)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — (hemothorax)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — (pneumothorax)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — (worsening of fibroids)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=1972)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 5 (5)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Foot Fracture (Injury, poisoning and procedural complications) | 2 (2)
Procedural Dizziness (Injury, poisoning and procedural complications) | 2 (2)
Procedural Pain (Injury, poisoning and procedural complications) | 2 (2)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Contusion (Injury, poisoning and procedural complications) | 1 (1)
Spinal Column Injury (Injury, poisoning and procedural complications) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1)
Paraesthesia (Injury, poisoning and procedural complications) | 10 (10)
Dizziness (Injury, poisoning and procedural complications) | 2 (2)
Migraine (Injury, poisoning and procedural complications) | 2 (2)
Neuropathy Peripheral (Injury, poisoning and procedural complications) | 1 (1)
Thoracic Outlet Syndrome (Injury, poisoning and procedural complications) | 1 (1)
Postoperative Wound Infection (Injury, poisoning and procedural complications) | 1 (2)
Cystitis (Injury, poisoning and procedural complications) | 1 (1)
Mastitis (Injury, poisoning and procedural complications) | 1 (1)
Urinary Tract Infection (Injury, poisoning and procedural complications) | 1 (1)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Warm (Skin and subcutaneous tissue disorders) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Food Allergy (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Influenza Like Illness (General disorders) | 1 (1)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast Discharge (Reproductive system and breast disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study are the property of Seno Medical Instruments, Inc. All publications (manuscripts, abstracts or other modes of presentation) must be submitted and reviewed and approved in writing by Seno Medical Instruments, Inc., in advance of submission. The over all study results will first be submitted as a primary paper.

DOCUMENTS (1):
  • Study Protocol (2015-10-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT01943916/Prot_000.pdf